CLINICAL TRIAL: NCT07373405
Title: Internet-based Interventions to Prevent the Development and Progression of Alcohol Use Disorders With and Without Internalizing and Externalizing Symptoms in Non-treatment Seekers: Protocol for a Nationwide Randomized Controlled Trial
Brief Title: Online Interventions to Prevent Alcohol Use Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20250010
Record Dates: First submitted 2025-12-10; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder (AUD)
Keywords: Alcohol Use Disorder; Internet-Based Interventions; Machine Learning; Non-treatment Seekers; Stepped-Care
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Internet-Based Brief Alcohol Intervention (Active Comparator)
  Interventions: Behavioral: Internet-Based Brief Alcohol Intervention
- Unguided Internet-Based Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Unguided Internet-Based Cognitive Behavioral Therapy
- Guided Internet-Based Cognitive Behavioral Therapy (Active Comparator)
  Interventions: Behavioral: Guided Internet-Based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Internet-Based Brief Alcohol Intervention — Brief Alcohol Intervention usually involves two components: assessing for hazardous alcohol use or AUD to identify problems early, and providing counselling. We are testing the effects of a digitalized version.
  Arms: Internet-Based Brief Alcohol Intervention
Behavioral: Unguided Internet-Based Cognitive Behavioral Therapy — Unguided Internet-based Cognitive Behavioral Therapy (iCBT) is a cost-effective intervention, where users complete structured, evidence-based CBT modules online without therapist involvement. The programs focus on teaching users techniques like identifying and challenging negative thoughts to manage - in this context - Alcohol Use Disorder symptoms.
  Arms: Unguided Internet-Based Cognitive Behavioral Therapy
Behavioral: Guided Internet-Based Cognitive Behavioral Therapy — Guided Internet-Based Cognitive Behavioral Therapy (iCBT) utilizes the structured, online delivery of CBT modules but adds regular, personalized support from a human therapist or trained coach. This human component typically involves checking assignments, providing motivational feedback, and tailoring advice to significantly boost user adherence and clinical outcomes.
  Arms: Guided Internet-Based Cognitive Behavioral Therapy

SUMMARY:
Background: Internet-based interventions can improve access to non-treatment-seeking populations, preventing the onset or progression of alcohol use disorder (AUD). Stepped-care guidelines for face-to-face AUD interventions recommend internet-based Brief Intervention (iBI) or unguided Cognitive Behavioural Therapy (iCBT) for no or mild AUD, and guided iCBT for moderate to severe AUD. However, no large-scale superiority trial has compared the effectiveness of these interventions among non-treatment-seeking individuals across the full spectrum of problematic alcohol use.

Aims: 1) Compare the effectiveness of iBI, unguided, and guided iCBT in reducing alcohol consumption in non-treatment-seeking individuals with sub-threshold or full AUD; 2) develop models via machine learning for personalized AUD prevention and progression management.

Methods: A nationwide sample of 3519 individuals will be stratified by sub-threshold/mild AUD and moderate/severe AUD and randomized to: 1) online assessment (OA)+ iBI; 2) OA+ unguided iCBT; or 3) OA+ guided iCBT. The iCBT sessions will address problematic alcohol use and co-occuring externalizing and internalizing psychiatric symptoms. Data will be collected from OA, interventions, and Danish registries at baseline and 3-, 6-, 12-, and 24-month follow-ups, with registry follow-up over 10 years.

Perspectives: Findings will compare stepped-care and machine learning-driven personalized approaches to inform guidelines for non-treatment-seeking populations. Internet-based assessment and interventions support continuous data collection, enabling ongoing improvements and personalized prevention. This large-scale dissemination targeting non-treatment-seeking populations across the full spectrum of problematic alcohol use will pave the way for future initiatives and may refine prevention strategies if the stepped-care model proves insufficient for this group.

Key words: Alcohol Use Disorder, Internet-Based Interventions, Machine Learning, Non-treatment Seekers, Stepped-Care

ELIGIBILITY:
Inclusion Criteria:

* Signing written informed consent
* Being aged ≥ 18 years
* Being a Danish resident and fluent in Danish
* Having at least weekly access to a computer or mobile phone with internet
* Having at least hazardous alcohol use, corresponding to an AUDIT cut-off score of ≥ 8/6 for men/women (no upper limit on the AUDIT score, as the alternative is no preventive intervention)

Exclusion Criteria:

* Receiving other psychological treatment
* Being suicidal or having severe comorbid psychiatric disorders (e.g., psychotic disorders).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3519 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Quantity-Frequency-Variability Index | From enrollment to 24 months.
  Alcohol consumption will be assessed using the Quantity-Frequency-Variability index, a quantity-frequency measure capturing drinking patterns over the past 7 and 30 days. The Quantity-Frequency-Variability index provides estimates of the number of drinking days, the number of drinks per drinking day, and the number of heavy drinking days (≥ 5 standard units of alcohol [SUA]). These measures are listed separately as distinct primary outcome measures.
Quantity-Frequency-Variability Index: Alcohol Frequency | From enrollment to 24 months.
  Measured using the Quantity-Frequency-Variability Index. Participants report the number of days they consumed alcohol in the past 7 and 30 days. Higher values indicate more frequent drinking.
Quantity-Frequency-Variability Index: Alcohol Quantity | From enrollment to 24 months.
  Measured using the Quantity-Frequency-Variability Index. Participants report the average number of standard units of alcohol (SUA) consumed on a typical drinking day in the past 30 days. Higher values indicate higher consumption per occasion.
Quantity-Frequency-Variability Index: Alcohol Variability | From enrollment to 24 months.
  Measured using the Quantity-Frequency-Variability Index. Participants report the number of days they consumed ≥ 5 standard units of alcohol (SUA) in the past 7 and 30 days. This captures the variability and pattern of drinking.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire Adapted to Internet-Based Interventions | Assessed at the 3-month follow-up assessment.
  The Client Satisfaction Questionnaire Adapted to Internet-Based Interventions includes 8 items measuring global satisfaction with web-based interventions. Each item is rated on a 4-point Likert scale ranging from 1 (does not apply to me) to 4 (does totally apply to me). The minimum score is 8 and the maximum score is 32. Higher scores indicate higher satisfaction.
System Usability Scale | Assessed at the 3-month follow-up assessment.
  The 10-item System Usability Scale will be used to measure subjective usability of internet-based interventions. The items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). The minimum score is 0 and the maximum score is 100. Higher scores indicate better usability.
Readiness-to-Change Questionnaire - Treatment Version | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  The Readiness-to-Change Questionnaire - Treatment Version is a 12-item measure designed to assess the respondent's stated intentions regarding changing their drinking behaviour. It includes three subscales representing different stages of change: (1) Pre-contemplation, (2) Contemplation, and (3) Action. Each subscale consists of four items, and responses are rated on a 5-point Likert Scale ranging from -2 (strongly disagree) to +2 (strongly agree). Total scores can range from -24 to +24. Higher scores on a specific subscale indicate greater alignment with that stage of change.
Alcohol Use Disorders Identification Test | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  The Alcohol Use Disorders Identification Test consists of 10 items assessing alcohol consumption, drinking behaviours, and alcohol-related problems. Items 1 to 8 are scored 0, 1, 2, 3 or 4, while items 9 and 10 are scored 0, 2 or 4. The total score can range from 0 to 40, with 0 indicating an abstainer who has never experienced any alcohol-related problems. In the study, only individuals who score ≥8 for men and ≥6 for women will be included, as scores from 1 to 7 for men and 1 to 5 for women suggest low-risk alcohol consumption according to WHO guidelines. Scores of 8 to 15 for men and 6 to 13 for women indicate hazardous or harmful alcohol consumption, while scores above 15 for men and above 13 for women suggest the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
Drug Use Disorders Identification Test | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  The Drug Use Disorders Identification Test consists of 11 items assessing drug use patterns and drug-related problems (excluding alcohol). Items 1 to 9 are scored 0, 1, 2, 3 or 4, while items 10 and 11 and are scored 0, 2 or 4. The total possible score ranges from 0 to 44, with higher scores reflecting higher drug dependence. A score of 6 for men and 2 for women indicates drug-related problems or harmful drug consumption, while a score of greater than 24 for both sexes suggests probable dependence on one or more drugs.
EuroQol five-dimensions-five-levels: Index Value | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  The EuroQol five-dimensions-five-levels assesses quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression, with five levels of severity for each (no problems, slight problems, moderate problems, severe problems, or extreme problems). The health state profile is converted into a single index value using the Danish value set (Jensen et al., 2023). In this context, the maximum score is 1.0, while the minimum score is -0.757. Higher scores indicates higher quality of life.
EuroQol five-dimensions-five-levels: Visual Analogue Scale | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  Participants rate their overall health on a vertical visual analogue scale. The scales ranges from 0 to 100. Higher scores indicate greater overall health perception.
Brief Symptom Inventory 18 | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  The Brief Symptom Inventory 18 is an 18-item questionnaire designed to assess psychological distress. Each item describes a symptom, and respondents rate the extent to which they have been bothered by the symptom over the past week on a 5-point scale, ranging from 0 (not at all) to 4 (extremely). Scores for all items are summarized on the Global Severity Index. The minimum score is 0 and the maximum score is 72. Higher scores indicate higher levels of psychological distress.
Buss-Perry Aggression Questionnaire - Short-Form | Assessed at baseline and at 3, 6, 12, and 24 months follow-up.
  The 12-item Buss-Perry Aggression Questionnaire - Short-Form consists of four subscales measuring hostility, anger, and physical and verbal aggression. Each subscale consists of three items, and responses are rated on a 5-point Likert scale ranging from 1 (extremely unlike me) to 5 (extremely like me). The minimum score is 12 and the maximum score is 60. Higher scores indicate higher levels of aggression.
Negative Effects Questionnaire | Assessed at the 3-month follow-up assessment.
  The Negative Effects Questionnaire includes 20 items rated on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely), distinguishing between negative effects attributed to the intervention and those potentially caused by other factors. The minimum score is 0 and the maximum score is 80. Higher scores indicate a higher burden of negative effects.
Register Data: Danish Education and Income Statistics Registers | Will be collected for 10 years from enrollment.
  Information on highest achieved education, employment, and economy will be retrieved.
Register Data: Danish National Patient Register | Will be collected for 10 years from enrollment.
  Data on inpatient and outpatient Alcohol Use Disorder-related contacts, prior Alcohol Use Disorder treatment, and other comorbidities will be collected.
Register Data: National Alcohol Treatment Register | Will be collected for 10 years from enrollment.
  Data on Alcohol Use Disorder treatment duration and intensity, treatment retention and type of treatment conclusion (i.e., dropout or completion), and prior Alcohol Use Disorder treatment will be retrieved.
Register Data: National Register of Substance Abusers in treatment | Will be collected for 10 years from enrollment.
  Data on Alcohol Use Disorder treatment duration and intensity, treatment retention and type of treatment conclusion (i.e., dropout or completion), and prior Alcohol Use Disorder treatment will be retrieved.
Register Data: Danish Prescription Register | Will be collected for 10 years from enrollment.
  Data on prescription of pharmacological treatment targeting Alcohol Use Disorder (e.g. disulfiram, naltrexone) and number of released receipts will be retrieved.
Register Data: Psychiatric Central Research Register | Will be collected for 10 years from enrollment.
  Data on inpatient and outpatient Alcohol Use Disorder-related contacts, prior Alcohol Use Disorder treatment, and other comorbidities will be collected.
Register Data: Cause of Death Register | Will be collected for 10 years from enrollment.
  Data on the date and primary cause of death, including both internal and external causes (accident, suicide, or murder), will be retrieved.